CLINICAL TRIAL: NCT04259294
Title: The Effects of a Home-based Occupational Therapy Tele-rehabilitation Via Smartphones for Outpatients After Hip Fracture Surgery in Hong Kong: A Feasibility Randomized Controlled Study
Brief Title: The Effects of a Home-based Occupational Therapy Tele-rehabilitation for Outpatients After Hip Fracture Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Kenneth N. K. Fong, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HongKongPOLYU
Record Dates: First submitted 2020-01-09; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation group via mobile apps (Experimental): The experimental group will receive home-based treatment program through mobile apps
  Interventions: Behavioral: Caspar Telerehabilitation
- Control group via paper and pencil instructions (Active Comparator): The control group will receive treatment via written home program sheets
  Interventions: Behavioral: Caspar Telerehabilitation

INTERVENTIONS:
Behavioral: Caspar Telerehabilitation — The experimental group will receive home-based treatment program through mobile apps while control group will receive through a written home program sheets. The training contents will be equivalent, including trunk and lower limb strengthening and stretching, coordination, balance, and functional exercises that will be related to patients' daily living activities in their home.
  The frequency and duration of the home program will be compromised by both the therapist and the patient. The videos of the home program will be sent to patients' app in smartphone by the therapist in the experimental group. Patients will perform the exercises while watching the videos in the app. After each exercise will be done, patient's performance feedback will be captured by the smartphone and will be sent back to the case therapist each time through the app while those in the control group will record their performance in a log sheet given by the therapists.

SUMMARY:
The investigators will investigate the effects of a home-based occupational therapy telerehabilitation (TR) via smartphones in enhancing functional and motor performances, and fall efficacy, for outpatients receiving day hospital rehabilitation after hip fracture surgery.

This is a feasibility randomized controlled trial with two groups - experimental and comparison groups, involving older adults after hip fracture surgery within 12 weeks attending the Geriatric Day Hospital. Patients will be assessed at baseline, immediately post 3-weeks intervention, and follow-up after 3-weeks for motor performances, daily activities functioning and fall efficacy. The experimental group will receive home program using the use of Caspar Health e-system and a mobile app in smartphones, while the comparison group will receive paper-and-pencil instructions for the home program on weekly basis, for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of hip fracture
* Post-hip surgery within 12 weeks
* Aged 60 years old or above
* Medically stable
* With Abbreviated Mental Test scored 6 or above
* Having at least one functional limitation in the basic activities of daily living assessments

Exclusion Criteria:

* The hip fracture is the result of malignancy
* There is risk of falls due to postural hypotension
* Either patients or caregiver do not understand Cantonese, English or Mandarin instructions
* They do not use a smartphone
* They are unable to read the instructions on the screen of the smartphone because of visual difficulty

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Timed up and go test (TUG) | Measure assessing change between three time points (baseline, post 3-week intervention and follow-up after 3 weeks)
  It measures fall risk and progress in walking speed (Change from baseline at post 3-week intervention and follow-up after 3 weeks)
The Functional Reach Test (FR) | Measure assessing change between three time points (baseline, post 3-week intervention and follow-up after 3 weeks)
  It measures balance (Change from baseline at post 3-week intervention and follow-up after 3 weeks)
Muscle strength (MS) | Measure assessing change between three time points (baseline, post 3-week intervention and follow-up after 3 weeks)
  It will be measured using a force gauge on the strength of Quadriceps of both the affected and the non-affected legs (Change from baseline at post 3-week intervention and follow-up after 3 weeks)
The Pain Visual Analogue Scale (VAS) | Measure assessing change between three time points (baseline, post 3-week intervention and follow-up after 3 weeks)
  It measures pain intensity. It consists of a 100mm horizontal line anchored with two opposite labels, i.e. labelled at the left end as 'no pain' (0mm) and at the right end as 'very severe pain' (100mm). (Change from baseline at post 3-week intervention and follow-up after 3 weeks)

SECONDARY OUTCOMES:
The Hong Kong Chinese version of the Modified Barthel index (MBI) | Measure assessing change between three time points (baseline, post 3-week intervention and follow-up after 3 weeks)
  It measures performance in basic activities of daily living. The item scores range from '0', which indicates an inability to perform, to a maximum of '5, 10 or 15', which represents total independence. The total items score of 100 indicates complete independence in self-care performance. (Change from baseline at post 3-week intervention and follow-up after 3 weeks)
The Hong Kong Chinese version of the Lawton Instrumental Activities of Daily Living (IADL) | Measure assessing change between three time points (baseline, post 3-week intervention and follow-up after 3 weeks)
  It assesses nine domains of function skills (ability to use telephone, shopping, meal preparation, laundry, housekeeping, handyman work, and transportation, medication and money management) The item scores range from '0' which indicates an inability to perform, to a maximum of '2,3 or 4' which represents total independence (Change from baseline at post 3-week intervention and follow-up after 3 weeks)
The Fall Efficacy Scale (FES) | Measure assessing change between three time points (baseline, post 3-week intervention and follow-up after 3 weeks)
  FES is a questionnaire to assess the level of confidence when patient perform activities of daily living without fear of fall. FES is a ten-item test rated on a 10-point scale from not confident at all to completely confident (Change from baseline at post 3-week intervention and follow-up after 3 weeks)
The Morse Fall Scale (MFS) | Measure assessing change between three time points (baseline, post 3-week intervention and follow-up after 3 weeks)
  MFS predict the likelihood of falls. It consists of 6 variables: history of fall, the presence of a secondary diagnosis, the use of ambulatory aids, the administration of intravenous therapy, types of gait and mental status. MFS is rated as follows, 0: No risk for falls; <25: Low risk; 25-45: Moderate risk ; >45: High risk (Change from baseline at post 3-week intervention and follow-up after 3 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong